CLINICAL TRIAL: NCT00114127
Title: Duloxetine for Social Anxiety Disorder: Prediction of Long Term Outcome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Naomi M. Simon, Director, Center for Anxiety and Traumatic Stress Disorders, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2004-P-001384
Record Dates: First submitted 2005-06-13; First posted 2005-06-14 (Estimated); Results first posted 2012-06-07 (Estimated); Last update posted 2014-06-10 (Estimated); Status verified 2014-06

CONDITIONS: Anxiety Disorder
Keywords: social anxiety disorder; social phobia; duloxetine; serotonin norepinephrine reuptake inhibitor; SNRI; double blind
MeSH Terms: conditions — Anxiety Disorders; Phobia, Social | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (3):
- Duloxetine 60mg + Placebo for 18 Weeks (Placebo Comparator): In Phase 2 participants were randomized to 60mg Duloxetine + Placebo or 120mg Duloxetine.
  Interventions: Drug: Duloxetine; Drug: Placebo
- Duloxetine 120mg for 18 Weeks (Active Comparator): In Phase 2 participants were randomized to 60mg Duloxetine + Placebo or 120mg Duloxetine.
  Interventions: Drug: Duloxetine
- Duloxetine 60mg/day for 6 Weeks (Active Comparator): In Phase 1 all participants entered an open trial.
  Interventions: Drug: Duloxetine

INTERVENTIONS:
Drug: Duloxetine — 60 mg duloxetine 1x per day
  Other Names: Cymbalta
  Arms: Duloxetine 60mg + Placebo for 18 Weeks; Duloxetine 60mg/day for 6 Weeks
Drug: Duloxetine — 60 mg duloxetine 1x per day + 60mg duloxetine 1x per day
  Other Names: Cymbalta
  Arms: Duloxetine 120mg for 18 Weeks
Drug: Placebo — 60mg placebo 1x per day
  Arms: Duloxetine 60mg + Placebo for 18 Weeks

SUMMARY:
The purpose of this study is to examine the safety and efficacy of duloxetine for the treatment of social anxiety disorder.

DETAILED DESCRIPTION:
An expanding body of clinical experience and controlled trials has established the efficacy of serotonin selective reuptake inhibitors (SSRIs) and the serotonin norepinephrine reuptake inhibitor (SNRI) venlafaxine, for the treatment of social anxiety disorder, with paroxetine, sertraline and venlafaxine extended-release (XR), which are FDA approved for this indication. The newest SNRI, duloxetine, has been shown to be effective at doses of 60mg/day to 120mg/day for anxiety associated with depression, and is anticipated to be a broad spectrum agent for mood and anxiety disorders (Dunner, Goldstein, Mallinckrodt, Lu, & Detke, 2003). However, no data on the efficacy of duloxetine for Social Anxiety Disorder, nor guidance regarding time to response or predictors of response, is yet available. These questions are the focus of this proposal.

This is a two phase, 24-week research study in which participants who remain symptomatic at the end of one phase (6 weeks) enter into the next phase. In phase I, all participants receive 60mg/day of duloxetine (Cymbalta) for 6 weeks. Participants who continue to have anxiety symptoms will enter the 18-week Phase II, in which they continue taking 60 mg/day of duloxetine and they will also be randomly assigned (by chance, like a flip of a coin) to receive either an additional 60mg/day of duloxetine or placebo (contains no active medication).

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients > 18 years of age with a primary psychiatric diagnosis of generalized social anxiety disorder as defined by DSM-IV criteria and an LSAS score > 50.
* Physical examination, electrocardiogram, and laboratory findings without clinically significant abnormalities.
* Willingness and ability to comply with the requirements of the study protocol.

Exclusion Criteria:

* Patient has a history of intolerance or lack of response to a treatment trial of duloxetine at highest tolerated dose (<120mg/day).
* Patients with acute narrow angle glaucoma.
* Pregnant women, lactating women, and women of childbearing potential who are not using medically accepted forms of contraception (e.g., IUD, oral contraceptives, barrier devices, condoms and foam, or implanted progesterone rods stabilized for at least 3 months).
* Concurrent use of other psychotropic medications. Patients must discontinue regular benzodiazepine or antidepressant therapy at least one week (5 weeks for fluoxetine) prior to baseline. Concomitant beta-blockers are proscribed unless prescribed for a medical indication (e.g., hypertension, at a stable daily dose for > 1 month).
* Patients with a history of failure to satisfactorily respond to >2 prior adequate treatment trials.
* Significant personality dysfunction likely to interfere with study participation.
* Serious medical illness or instability for which hospitalization may be likely within the next year.
* Seizure disorders with the exception of a history of febrile seizures if they occurred during childhood, were isolated, and did not recur in adulthood.
* Concurrent psychotherapy initiated within 2 months of baseline is prohibited. Ongoing psychotherapy of any duration directed specifically toward treatment of the social anxiety disorder is excluded. Prohibited psychotherapy includes cognitive behavioral therapy or psychodynamic therapy that focuses on exploring specific, dynamic causes of the phobic symptomatology and provides skills for their management. General supportive individual, couples, or family therapy greater than 2 months duration is acceptable.
* Diagnosis of any of the following mental disorders as defined by the DSM-IV: a lifetime history of schizophrenia or any other psychosis, mental retardation, organic medical disorders or bipolar disorder; eating disorders in the past 6 months; alcohol or substance abuse in the past 3 months or dependence within the past 6 months.
* Entry of patients with major depression, dysthymia, panic disorder, generalized anxiety disorder, post-traumatic stress disorder or obsessive-compulsive disorder will be permitted if the social anxiety disorder is judged to be the predominant disorder, in order to increase accrual of a clinically relevant sample.
* Patients with significant suicidal ideation (MADRS item 10 score > 3) or who have enacted suicidal behaviors within 6 months prior to intake will be excluded from study participation and referred for appropriate clinical intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2004-06; Primary Completion 2008-11 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naomi M Simon, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- See also: Official Website for the Center for Anxiety and Traumatic Stress Disorders — http://www.mghanxiety.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Treatment seeking outpatients aged 18 years and older with a primary diagnosis of Generalized Social Anxiety Disorder (GSAD) were recruited by media advertisement.
Pre-assignment Details: Of the 39 participants who completed Phase I of this study, 28 moved on to Phase II.
  1 subject was lost to follow up between baseline and week 1.
Groups:
- Duloxetine 60mg/Day + Placebo for 18 Weeks (Phase 2): Participants who did not achieve remission at the end of Phase 1 entered Phase 2 and were randomized. 13 received 60mg duloxetine plus placebo for 18 additional weeks.
- Duloxetine 120mg/Day for 18 Weeks (Phase 2): Participants who did not achieve remission at the end of Phase 1 entered Phase 2 and were randomized. 15 received 120mg duloxetine for 18 additional weeks.
Period: Overall Study
Arm/Group | Duloxetine 60mg/Day + Placebo for 18 Weeks (Phase 2) | Duloxetine 120mg/Day for 18 Weeks (Phase 2)
Started | 13 | 15
Completed | 9 | 11
Not Completed | 4 | 4
Not completed — Adverse Event | 2 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Duloxetine 60mg/Day + Placebo for 18 Weeks(Phase 2): Participants who did not achieve remission at the end of Phase 1 entered Phase 2 and were randomized. 13 received 60mg duloxetine plus placebo for 18 additional weeks.
- Total: Total of all reporting groups
Arm/Group | Duloxetine 60mg/Day + Placebo for 18 Weeks(Phase 2) | Duloxetine 120mg/Day for 18 Weeks (Phase 2) | Total
Number analyzed (Participants) | 13 | 15 | 28
Age, Customized [Mean (Standard Deviation); unit: Years]
  Age Baseline | 36.6 (14.2) | 35.5 (11.6) | 36 (12.6)
Sex/Gender, Customized [Number; unit: Participants]
  Female | 7 | 4 | 11
  Male | 6 | 11 | 17
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 9 | 13 | 22
  Asian | 1 | 1 | 2
  Black | 1 | 1 | 2
  Alaskan Native | 1 | 0 | 1
  Native Hawaiian or Pacific Islander | 1 | 0 | 1
Educational status, college graduate [Number; unit: Participants]
  College Graduate | 10 | 7 | 17
  Not College Graduate | 3 | 8 | 11
Duration of illness, mean years (SD) [Mean (Standard Deviation); unit: Years] | 27.6 (17.0) | 20.1 (12.3) | 23.7 (14.9)
Age of onset, mean age [Mean (Standard Deviation); unit: Years] | 9.9 (3.3) | 13.9 (8.1) | 12.0 (6.46)
Current comorbidity, Major depressive disorder (MDD) [Number; unit: Participants]
  Comorbid MDD | 5 | 0 | 5
  No Comorbid MDD | 8 | 15 | 23
Current comorbidity, Dysthymia [Number; unit: Participants]
  Comorbid Dysthymia | 2 | 0 | 2
  No Comorbid Dysthymia | 11 | 15 | 26
Current comorbidity, Panic Disorder (PD) [Number; unit: Participants]
  Comorbid PD | 1 | 0 | 1
  No Comorbid PD | 12 | 15 | 27
Current comorbidity, Generalized anxiety disorder (GAD) [Number; unit: Participants]
  Comorbid GAD | 2 | 0 | 2
  No Comorbid GAD | 11 | 15 | 26
At least one concurrent mood or anxiety disorder [Number; unit: Participants]
  Concurrent mood or anxiety disorder | 7 | 1 | 8
  No concurrent mood or anxiety disorders | 6 | 14 | 20
Lifetime depression [Number; unit: Participants]
  Lifetime depression | 6 | 4 | 10
  No Lifetime depression | 7 | 11 | 18
Lifetime alcohol or substance abuse or dependence [Number; unit: Participants]
  Lifetime Alcohol/substance abuse/dependence | 3 | 3 | 6
  No Lifetime Alcohol/substance abuse/dependence | 10 | 12 | 22
Liebowitz Social Anxiety Scale (LSAS) [Mean (Standard Deviation); unit: LSAS Score] — The Liebowitz Social Anxiety Scale (LSAS; Liebowitz, 1987) is a 24-item scale that provides separate scores for fear and avoidance in social and performance situations with higher scores representing increased social anxiety (55-65 Moderate social phobia, 65-80 Marked social phobia, 80-95 Severe social phobia, Greater than 95 - Very severe social phobia). It is widely used in treatment studies of SAD. The instrument shows very good psychometric properties (Heimberg et al., 1999; Safren et al., 1999).
  Baseline collected for Phase 1 at week 0 and for Phase 2 at week 6.
  LSAS Score | 75.2 (6.90) | 74.1 (6.20) | 74.6 (4.52)
Clinical Global Impression-Severity (CGI-S) [Mean (Standard Deviation); unit: CGI-S Score] — The Clinician Global Impression-Severity Scale (CGI-S) is a clinician-rated instrument used to assess global severity of symptoms (Guy, 1976). The CGI ranges from 1 (normal, not at all ill) to 7 (among the most extremely ill patients).
  Baseline collected for Phase 1 at week 0 and for Phase 2 at week 6.
  CGI-S Score | 5.10 (0.43) | 4.93 (0.36) | 5.00 (0.27)
Clinical Global Impression-Improvement (CGI-I) [Mean (Standard Deviation); unit: CGI-I Score] — The Clinician Global Impression-Improvement Scale (CGI-I) is a clinician-rated instrument used to assess global improvement of symptoms (Guy, 1976). The CGI ranges from 1 (very much improved) to 7 (very much worse).
  Baseline CGI-I was not collected in Phase 1 as it is a measure of improvement. Baseline CGI-I was collected in Phase 2 because patients were transitioning from week 6 to 7.
  CGI-I Score | 3.25 (0.97) | 3.36 (1.22) | 3.31 (1.09)
Montgomery Asberg Depression Rating Scale (MADRS) [Mean (Standard Deviation); unit: MADRS Score] — MADRS; Montgomery & Asberg, 1979. The MADRS is designed to measure the overall severity of depressive symptoms and has demonstrated good reliability and sensitivity to change with treatment. It includes 10 items and uses a 0-6 severity scale with higher scores indicating increasing depressive symptoms. Ratings can be added to form an overall score (range 0 to 60); no weights are used. Cut-off points include: 0 to 6 - symptom absent, 7 to 19 - mild depression, 30 to 34 - moderate, 35 to 60 - severe depression.
  Baseline MADRS only collected in Phase 2 at week 6.
  MADRS Score | 8.08 (5.00) | 10.3 (7.79) | 9.17 (6.60)
Sheehan Disability Scale (SDS) [Mean (Standard Deviation); unit: SDS Score] — The SDS is a brief self-report questionnaire that was developed to assess functional impairment in three inter-related domains; work/school, social and family life. The patient rates the extent to which work/school, social and family responsibilities are impaired by his/her symptoms on a 10 point visual analog scale. The three items are summed into a single dimension measure of global function impairment that ranges from 0 (unimpaired) to 30 (highly impaired).
  Baseline SDS only collected in Phase 2 at week 6.
  SDS Score | 11.2 (6.06) | 14.1 (5.52) | 12.9 (5.71)
Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q) [Mean (Standard Deviation); unit: Q-LES-Q Score] — Q-LES-Q; Endicott et al., 1993. This questionnaire rates 16 aspects of quality of life, including physical health, mood, activities of daily living, and overall life satisfaction. The scoring of the Q-LES-Q-SF involves summing only the first 14 items to yield a raw total score. The last two items are not included in the total score but are standalone items. The raw total score ranges from 14 to 70, with higher scores indicating higher satisfaction with quality of life.
  Baseline QLESQ only collected in Phase 2 at week 6.
  Q-LES-Q Score | 49.1 (8.83) | 46.2 (9.47) | 47.5 (9.12)
Liebowitz Self-Rated Disability Scale (LSDSR) [Mean (Standard Deviation); unit: LSDSR Score] — The Liebowitz Social Anxiety Scale (LSAS; Liebowitz, 1987) is a 24-item scale that provides separate scores for fear and avoidance in social and performance situations with higher scores representing increased social anxiety. The LSAS contains three total scores: 1) total fear score (0-72), 2) total avoidance score(0-72), 3) and total overall score (0-144). Suggested interpretations: 55-65 Moderate social phobia, 65-80 Marked social phobia, 80-95 Severe social phobia, Greater than 95 - Very severe social phobia.
  Baseline was only collected for Phase 2 at week 6
  LSDSR Score | 7.58 (6.43) | 10.0 (5.41) | 8.79 (5.83)

OUTCOME MEASURES:

1. Primary Outcome: Anxiety Symptoms as Assessed by Liebowitz Social Anxiety Scale
Description: The Liebowitz Social Anxiety Scale (LSAS; Liebowitz, 1987) is a 24-item scale that provides separate scores for fear and avoidance in social and performance situations with higher scores representing increased social anxiety. The LSAS contains three total scores: 1) total fear score (0-72), 2) total avoidance score(0-72), 3) and total overall score (0-144). Suggested interpretations: 55-65 Moderate social phobia, 65-80 Marked social phobia, 80-95 Severe social phobia, Greater than 95 - Very severe social phobia.
Time Frame: 6 months
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | Duloxetine 60mg/Day + Placebo for 18 Weeks (Phase 2) | Duloxetine 120mg/Day for 18 Weeks (Phase 2)
Number analyzed (Participants) | 13 | 15
Scores on a scale | 67.9 (7.60) | 53.7 (7.90)
Statistical Analysis 1: Comparison: Duloxetine 60mg/Day + Placebo for 18 Weeks (Phase 2) vs Duloxetine 120mg/Day for 18 Weeks (Phase 2); Test type: Superiority or Other; p < 0.132, t-test, 2 sided

2. Secondary Outcome: CGI-S
Description: The Clinician Global Impression-Severity Scale (CGI-S) is a clinician-rated instrument used to assess global severity of symptoms (Guy, 1976). The CGI ranges from 1 (normal, not at all ill) to 7 (among the most extremely ill patients).
  Baseline collected for Phase 1 at week 0 and for Phase 2 at week 6.
Time Frame: 6 months
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | Duloxetine 60mg/Day + Placebo for 18 Weeks (Phase 2) | Duloxetine 120mg/Day for 18 Weeks (Phase 2)
Number analyzed (Participants) | 13 | 15
Scores on a scale | 4.42 (0.48) | 3.60 (0.57)
Statistical Analysis 1: Comparison: Duloxetine 60mg/Day + Placebo for 18 Weeks (Phase 2) vs Duloxetine 120mg/Day for 18 Weeks (Phase 2); Test type: Superiority or Other; p < .292, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Duloxetine 60mg/Day + Placebo for 18 Weeks (Phase 2) | Duloxetine 120mg/Day for 18 Weeks (Phase 2)
Serious Adverse Events (participants affected / at risk) | 2/13 | 0/15
Other Adverse Events (participants affected / at risk) | 0/13 | 2/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Duloxetine 60mg/Day + Placebo for 18 Weeks (Phase 2) (N=13) | Duloxetine 120mg/Day for 18 Weeks (Phase 2) (N=15)
Elevated Liver Function Tests (General disorders) | 1 (1) | 0 (0) — The elevated LFTs were later diagnosed by primary care physician on evaluation as unrelated to study medication and a result of rhabdomyolysis from a week of intensive weight lifting and exercises.
Study medication overdose (General disorders) | 1 (1) | 0 (0) — The study medication overdose was in the context of alcohol use and suicidal ideation and had no medical consequences: this was deemed possibly related to duloxetine and the participant was transferred to clinical care.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Duloxetine 60mg/Day + Placebo for 18 Weeks (Phase 2) (N=13) | Duloxetine 120mg/Day for 18 Weeks (Phase 2) (N=15)
Sedation and other side effects (General disorders) | 0 (0) | 1 (1)
Increased drinking (General disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Open-label in phase Phase 1; Limited power due to small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No